CLINICAL TRIAL: NCT00244140
Title: Ultravist 370 Milligrams of Iodine Per Milliliter (mg I/mL): Safety and Efficacy in Computed Tomography of Head and Body
Brief Title: Ultravist: Safety and Efficacy in Computed Tomography of Head and Body
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 91462; 309660 (Other: company internal)
Record Dates: First submitted 2005-10-24; First posted 2005-10-26 (Estimated); Results first posted 2009-07-20 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Computed Tomography; Diagnostic Imaging
Keywords: Ultravist 370; CECT; CT Scan
MeSH Terms: interventions — iopromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iopromide 370 mg I/mL (Experimental): Iopromide (Ultravist 370 mg I/mL) administered intravenously
  Interventions: Drug: Iopromide 370 mg I/mL
- Iopromide 300 mg I/mL (Experimental): Iopromide (Ultravist 300 mg I/mL) administered intravenously
  Interventions: Drug: Iopromide 300 mg I/mL

INTERVENTIONS:
Drug: Iopromide 370 mg I/mL — Iopromide (Ultravist 370 mg I/mL) administered intravenously
  Arms: Iopromide 370 mg I/mL
Drug: Iopromide 300 mg I/mL — Iopromide (Ultravist 300 mg I/mL) administered intravenously
  Arms: Iopromide 300 mg I/mL

SUMMARY:
This is a research study involving the use of a contrast agent called Ultravist Injection. Ultravist, the study drug, is used to improve the pictures obtained using computed tomography (CT). Ultravist acts like a dye to make CT pictures brighter and easier to read. In the case of this study, it will be injected into a vein in the patient's arm; from there, it travels through the blood stream and to the areas to be examined. CT scans will then be taken of the patient's head and/or body as ordered by his/her physician.

Phase IIIb Study to Document the Safety and Efficacy of Ultravist 370 mg I/ml, When Administered Intravenously, in Volumes up to 162.2 ml, for Clinically Indicated Contrast Enhanced Computed Tomography (CECT) of the Head and/or Body

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.

Bayer HealthCare Pharmaceuticals, Inc. is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years old and clinically indicated for a contrast-enhanced CT of the head or body.

Exclusion Criteria:

* Patients that are less than 18 years old and do not have a clinical indication for a contrast-enhanced CT of the head or body.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2005-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- United States (14):
  - Tucson, Arizona
  - Miami, Florida
  - Tallahassee, Florida
  - Atlanta, Georgia
  - Evanston, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - New York, New York
  - Stony Brook, New York
  - Cleveland, Ohio
  - Danville, Pennsylvania
  - Charleston, South Carolina
- Colombia (2):
  - Medellín, Antioquia
  - Bogotá
- India (2):
  - Mumbai-400026
  - Tamil Nadu
- South Korea (2):
  - Seoul, Seoul Teugbyeolsi
  - Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was 21 Oct 2005 to 11 Apr 2008.
Pre-assignment Details: 437 subjects were screened; 2 subjects were screen failures because of not meeting inclusion criteria and/or meeting exclusion criteria; 435 subjects were enrolled; 1 enrolled subject withdrew consent before receiving study drug; 434 subjects received study drug and were included in the safety analysis set.
Period: Overall Study
Arm/Group | Iopromide 370 mg I/mL | Iopromide 300 mg I/mL
Started | 412 | 22
Completed | 412 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iopromide 370 mg I/mL | Iopromide 300 mg I/mL | Total
Number analyzed (Participants) | 412 | 22 | 434
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (15.15) | 56.5 (14.54) | 52.1 (15.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 16 | 207
  Male | 221 | 6 | 227

OUTCOME MEASURES:

1. Primary Outcome: The Quality of Visualization of the Contrast-Enhanced Computed Tomography (CECT) Images, Based on the Blinded Readers' Assessment.
Description: A subjective assessment of the 'Quality of Image' (QOI) by 3 blinded readers (BR). QOI-Grades used: Excellent - Good - Poor.
Time Frame: post administration assessment of study images
Population: The primary efficacy analysis used the Full Analysis Set (FAS), which consisted of the subjects who received any amount of iopromide regardless of any protocol deviation, excluding the sample subjects and subjects who did not have CT images. In the FAS, 402 subjects were included.
Measure: Number; unit: Number of participants in QOI grade
Arm/Group | Iopromide 370 mg I/mL | Iopromide 300 mg I/mL
Number analyzed (Participants) | 382 | 20
Number of participants in QOI grade
  Excellent + Good (blinded reader 1) | 366 | 17
  Poor (blinded reader 1) | 16 | 3
  Excellent + Good (blinded reader 2) | 368 | 19
  Poor (blinded reader 2) | 14 | 1
  Excellent + Good (blinded reader 3) | 376 | 15
  Poor (blinded reader 3) | 6 | 5
Statistical Analysis 1: Comparison: Iopromide 370 mg I/mL; Study was uncontrolled - No comparison between groups. The 95% Confidence Interval (CI) were calculated for each of the 3 blinded readers separately. This analysis refers to the assessment of blinded reader 1 (BR1); Test type: Superiority or Other; Percent Images Rated Good/Excellent: BR1 = 95.8, 95% CI [93.3 to 97.6]
Statistical Analysis 2: Comparison: Iopromide 370 mg I/mL; Study was uncontrolled - No comparison between groups. The 95% Confidence Interval (CI) were calculated for each of the 3 blinded readers separately. This analysis refers to the assessment of blinded reader 2 (BR2); Test type: Superiority or Other; Percent Images Rated Good/Excellent: BR2 = 96.3, 95% CI [93.9 to 98.0]
Statistical Analysis 3: Comparison: Iopromide 370 mg I/mL; Study was uncontrolled - No comparison between groups. The 95% Confidence Interval (CI) were calculated for each of the 3 blinded readers separately. This analysis refers to the assessment of blinded reader 3 (BR3); Test type: Superiority or Other; Percent Images Rated Good/Excellent: BR3 = 98.4, 95% CI [96.6 to 99.4]

2. Secondary Outcome: The Ability of the Investigator to Make a Diagnosis Based on the CECT Images
Description: The number of participants with diagnostic CECTs as assessed by the investigators.
Time Frame: post administration assessment of study images
Population: as for outcome 1
Measure: Number; unit: Number of diagnostic CECTs
Arm/Group | Iopromide 370 mg I/mL | Iopromide 300 mg I/mL
Number analyzed (Participants) | 382 | 20
Number of diagnostic CECTs
  No | 1 | 0
  Not applicable | 0 | 0
  Yes | 381 | 20
Statistical Analysis 1: Comparison: Iopromide 370 mg I/mL; Test type: Superiority or Other; Percent Images Rated Yes = 99.7, 95% CI [98.6 to 100.0]

3. Secondary Outcome: The Quality of Visualization of the Contrast-Enhanced Computed Tomography (CECT) Images, Based on the Investigators' Assessment.
Description: A subjective assessment of the 'Quality of Image' (QOI) by the investigators. QOI-Grades used: Excellent - Good - Poor.
Time Frame: post administration assessment of study images
Population: as for outcome 1
Measure: Number; unit: Number of participants in QOI grade
Arm/Group | Iopromide 370 mg I/mL | Iopromide 300 mg I/mL
Number analyzed (Participants) | 382 | 20
Number of participants in QOI grade
  Excellent + Good | 380 | 20
  Poor | 2 | 0
Statistical Analysis 1: Comparison: Iopromide 370 mg I/mL; Test type: Superiority or Other; Percent Images Rated Good/Excellent = 99.5, 95% CI [98.1 to 99.9]

4. Secondary Outcome: The Ability of the Blinded Readers to Make a Diagnosis Based on the CECT Images
Description: The number of participants with diagnostic CECTs as assessed by the 3 blinded readers.
Time Frame: post administration assessment of study images
Population: as for outcome 1
Measure: Number; unit: Number of diagnostic CECTs
Arm/Group | Iopromide 370 mg I/mL | Iopromide 300 mg I/mL
Number analyzed (Participants) | 382 | 20
Number of diagnostic CECTs
  No (blinded reader 1) | 6 | 2
  Not applicable (blinded reader 1) | 0 | 0
  Yes (blinded reader 1) | 376 | 18
  No (blinded reader 2) | 0 | 0
  Not applicable (blinded reader 2) | 0 | 0
  Yes (blinded reader 2) | 382 | 20
  No (blinded reader 3) | 0 | 0
  Not applicable (blinded reader 3) | 1 | 0
  Yes (blinded reader 3) | 381 | 20
Statistical Analysis 1: Comparison: Iopromide 370 mg I/mL; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Percent Images Rated Yes: BR1 = 98.4, 95% CI [96.6 to 99.4]
Statistical Analysis 2: Comparison: Iopromide 370 mg I/mL; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Percent Images Rated Yes: BR2 = 100.0, 95% CI [99.0 to 100.0]
Statistical Analysis 3: Comparison: Iopromide 370 mg I/mL; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Percent Images Rated Yes: BR3 = 99.7, 95% CI [98.6 to 100.0]

ADVERSE EVENTS:
Arm/Group | Iopromide 370 mg I/mL | Iopromide 300 mg I/mL
Serious Adverse Events (participants affected / at risk) | 2/412 | 0/22
Other Adverse Events (participants affected / at risk) | 32/412 | 1/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iopromide 370 mg I/mL (N=412) | Iopromide 300 mg I/mL (N=22)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iopromide 370 mg I/mL (N=412) | Iopromide 300 mg I/mL (N=22)
Nausea (Gastrointestinal disorders) | 6 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 5 | 0
Feeling Hot (General disorders) | 4 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Haemoglobin increased (Investigations) | 2 | 0
White blood cell count increased (Investigations) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less